CLINICAL TRIAL: NCT05421780
Title: Impact of Brewer's Spent Grain (BSG) and Bio-transformed BSG Biscuits on Post-prandial Glycaemic Controlling Effects in Singapore Adults With Metabolic Syndrome
Brief Title: Post-prandial Glycaemic Controlling Effects of BSG in Singapore Adults With Metabolic Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University of Singapore (Other)
Collaborators: Ministry of Education, Singapore (Other Government)
Responsible Party: Principal Investigator, Jung Eun Kim, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: S16
Record Dates: First submitted 2022-05-30; First posted 2022-06-16 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Metabolic Syndrome; Diabetes; Diet Modification
Keywords: Metabolic Syndrome; middle-aged and older adults; Post-prandial Glycaemic response; bio-transformed food
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control biscuits group (Placebo Comparator): For each MTT, subjects are to consume 90 g control biscuits as their breakfast within 15 mins.
  Interventions: Dietary Supplement: control biscuits
- autoclaved BSG-containing group (Experimental): For each MTT, subjects are to consume 90 g autoclaved BSG-containing biscuits as their breakfast within 15 mins.
  Interventions: Dietary Supplement: autoclaved BSG-containing biscuits
- bio-transformed BSG-containing group (Experimental): For each MTT, subjects are to consume 90 g bio-transformed BSG-containing biscuits as their breakfast within 15 mins.
  Interventions: Dietary Supplement: bio-transformed BSG-containing biscuits

INTERVENTIONS:
Dietary Supplement: autoclaved BSG-containing biscuits — Consumption of autoclaved BSG-containing biscuits as breakfast.
  Arms: autoclaved BSG-containing group
Dietary Supplement: bio-transformed BSG-containing biscuits — Consumption of bio-transformed BSG-containing biscuits as breakfast.
  Arms: bio-transformed BSG-containing group
Dietary Supplement: control biscuits — Consumption of plain biscuits as breakfast.
  Arms: Control biscuits group

SUMMARY:
The purpose of this study is to assess the glycaemic controlling effects of BSG and bio-transformed BSG-containing biscuits in Singapore adults with MetS. The investigators hypothesized that consumption of BSG and bio-transformed BSG containing biscuit will improve glycaemic control.

DETAILED DESCRIPTION:
This is a double-blind, randomised, crossover experiment. During the 3-week, 19 subjects will participate in a 3 meal tolerance test (MTT). During each MTT session, all subjects are required to consume 90 g biscuits (either control, autoclaved BSG or bio-transformed BSG biscuits) and monitored over a period of 240 minutes. All three types of biscuits will be consumed at a randomised sequence during this 3-week period. Post-prandial blood glucose, insulin, lipid and amino acid responses, breath analysis, body composition, blood pressure, appetite assessment, and any other glycaemic biomarkers will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants, aged 35-85 years old
* English-literate and able to give informed consent in English
* Willing to follow the study procedures
* Meet any 3 of the 5 following NCEP-ATP III MetS criteria: waist circumference > 102 cm (male), > 88 cm (female) (For Asian population: Waist circumference > 90 cm (male), > 80 cm (female)); fasting glucose concentration ≥ 100 mg/dL or on medication; triglyceride ≥ 150 mg/dL or on medication; high density lipoprotein cholesterol (HDL) < 40 mg/dL (male), < 50 mg/dL (female); systolic or diastolic blood pressure > 130/85 mmHg or on medication);

Exclusion Criteria:

* Significant change in weight (≥ 3 kg body weight) during the past 3 months
* Allergy to barley, wheat, corn, egg, or other ingredients found inside the biscuits.
* Acute illness at the study baseline
* Exercising vigorously* over the past 3 months. *Defined as having > 6 metabolic equivalents of exercise daily; approximately 20 mins of moderate intensity exercise (e.g. slow jogging) a day
* Following any restricted diet (e.g. vegetarian)
* Smoking
* Have a daily intake of more than 2 alcoholic drinks per day
* Taking dietary supplements or food which may impact the outcome of interests (e.g. fermented foods, probiotic supplement etc.)
* Consumption of antibiotics over past 3 months.
* Pregnant, lactating, or planning pregnancy in the next 6 months
* Insufficient venous access to allow the blood collection
* Prescribed and taking antihypertensive/cholesterol-lowering/ type-2 diabetic medication which started less than 3 years prior to the intervention participation
* High current intake of fibre* from brown rice or wholemeal products. *High, moderate or low intake taken as ≥ 6 servings, 4 - 5 servings, and ≤ 3 servings daily respectively based on My Healthy Plate guidelines
* High current intake of fibre* from vegetables. * High, moderate or low intake taken as ≥ 2 servings, 2 servings, and ≤ 1 serving respectively based on My Healthy Plate guidelines

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Change in blood glucose concentration | Every week (week 1, week 2 and week 3)
  Glucose concentration in the blood will be measured
Change in blood insulin concentration | Every week (week 1, week 2 and week 3)
  Insulin concentration in the blood will be measured
Change in blood triglyceride concentration | Every week (week 1, week 2 and week 3)
  Triglyceride concentration in the blood will be measured
Change in blood cholesterol concentration | Every week (week 1, week 2 and week 3)
  Total cholesterol concentration in the blood will be measured
Change in blood Low-density Lipoprotein-cholesterol (LDL) concentration | Every week (week 1, week 2 and week 3)
  Low-density Lipoprotein-cholesterol concentration in the blood will be measured
Change in High-density Lipoprotein-cholesterol (HDL) concentration | Every week (week 1, week 2 and week 3)
  High-density Lipoprotein-cholesterol concentration in the blood will be measured
Change in blood amino acid concentration | Every week (week 1, week 2 and week 3)
  Amino acid concentration in the blood will be measured

SECONDARY OUTCOMES:
Change in appetite assessed by visual analogue scale | Every week (week 1, week 2 and week 3)
  Visual analogue scale will be used to assess appetite.
Change in breath CH4 and H2 concentrations | Every week (week 1, week 2 and week 3)
  CH4 and H2 concentrations will be measured by breath analyzer
Change in weight and height | Every week (week 1, week 2 and week 3)
  Weight (in kilograms) and height (in meters) will be combined to report BMI in kg/m^2
Change in waist circumference | Every week (week 1, week 2 and week 3)
  Waist circumference (in cm) will be measured
Change in blood pressure | Every week (week 1, week 2 and week 3)
  Systolic and diastolic blood pressure (in mmHg) will be measured by a blood pressure monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Jung Eun Kim, Principal Investigator — Food Science and technology, Faculty of Science, National University of Singapore
Locations (1):
- Yujing Xu, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Electronic copies of the data with identifiable participant information will be kept on a secure website with access limited to Dr. Kim and Dr. Kim's research staff. All data will be de-identified prior to statistical analyses.